CLINICAL TRIAL: NCT01326455
Title: Caring for the Radial Artery Post-angiogram: A Pilot Study on a Comparison of Three Methods of Compression
Brief Title: Caring for the Radial Artery Post-angiogram
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: Pro00005016
Record Dates: First submitted 2011-03-29; First posted 2011-03-30 (Estimated); Results first posted 2022-09-28 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2011-09

CONDITIONS: Transradial Angiogram
Keywords: transradial; angiogram; device; Care of the radial artery post transradial angiogram

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Terumo Control (Other)
  Interventions: Device: Terumo TR wristband
- Terumo Fast Release (Active Comparator)
  Interventions: Device: Terumo TR wristband
- Clo-Sur P.A.D. (Active Comparator)
  Interventions: Device: Clo-Sur-P.A.D.

INTERVENTIONS:
Device: Terumo TR wristband — A transparent unilateral compression device which is secured to the wrist via strap with velcro. The portion with the deflated 18cc balloon is placed directly over the puncture site. This balloon is inflated immediately after the catheter is removed and the balloon is inflated until bleeding visibly stops, with generally 9-18cc of air.
  First deflation of 3cc of air occurred 1 hour after inflation. Deflations occurred every 15 minutes unless bleeding was noted. If bleeding was noted, balloon was reinflated (1-3cc of air) until bleeding stopped. Next deflation occurred 30 minutes later, at which point regular 15 minutes deflations occurred if no bleeding noted. Band was removed 1 hour after final deflation.
  Arms: Terumo Control
Device: Terumo TR wristband — A transparent unilateral compression device which is secured to the wrist via strap with velcro. The portion with the deflated 18cc balloon is placed directly over the puncture site. This balloon is inflated immediately after the catheter is removed and the balloon is inflated until bleeding visibly stops, with generally 9-18cc of air.
  First balloon deflation of 3cc of air occurred 15 minutes after initial inflation. Deflations occurred every 15 minutes unless bleeding was noted. If active bleeding was noted, the balloon was re-inflated (1-3cc) until bleeding stopped. The next deflation occurred 15 minutes later. If no bleeding occurred, deflations continued every 15 minutes until the balloon was completely deflated. The band was removed 15 minutes after final deflation.
  Arms: Terumo Fast Release
Device: Clo-Sur-P.A.D. — A hydrophilic dressing has a high affinity for water, and absorbs and controls body fluid. The positively charged 4x4 centimetre pad reacts with the neuraminic acid residue on red blood cells causing agglutination of the cells. The Clo-Sur P.A.D. works outside of the clotting cascade.
  The radial catheter was removed and occlusive pressure applied on the radial artery. Pressure was released just until bleeding noted & the pad was applied with approximately 5 minutes of manual compression. The pad was assessed every 15 minutes for 90 minutes to ensure hemostasis. The pad was removed on post-CATH day 1.
  Arms: Clo-Sur P.A.D.

SUMMARY:
The purpose of this pilot study was to compare two devices and three methods for achieving hemostasis after a transradial angiogram while assessing vascular complications and time endpoints. The heart has traditionally been accessed through the femoral artery. However, in the last 20 years, the radial artery has gained more popularity among physicians and patients, thereby offering an alternative to the femoral approach. Various methods of applying compression to the radial puncture site have been used, but no research has been done to show what best practice is. In this case, best practice would be the most effective way of getting hemostasis while limiting complications and ensuring the efficient use of nursing and medical resources. It is hypothesized that statistically significant differences are seen in time to discharge in the fast-release Terumo and Clo-Sur P.A.D. groups, as compared with the control Terumo group, without increasing vascular complications.

ELIGIBILITY:
Inclusion Criteria:

* nonemergent
* outpatient

Exclusion Criteria:

* inpatients
* emergency patients
* booked angioplasty patients
* cognitive impairment
* those in whom the approach was initiated but aborted due to inability to puncture the radial artery

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2009-05; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Colleen Norris, PhD, Principal Investigator — University of Alberta

REFERENCES:
- [Background] Fech JC, Welsh R, Hegadoren K, Norris CM. Caring for the radial artery post-angiogram: a pilot study on a comparison of three methods of compression. Eur J Cardiovasc Nurs. 2012 Mar;11(1):44-50. doi: 10.1177/1474515111429656. Epub 2012 Jan 11. PMID 22357780

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The pilot study was set in one Cardiac Cath Lab and Recovery room. The sample was one of convenience. The goal was for 75 people to participate, 25 per group. The individuals targeted were those having an angiogram done on a non-emergent, outpatient basis. Recruitment took place from May 2009 until March 2010.
Pre-assignment Details: Participants were enrolled prior to the angiogram. Those patients in whom the transradial approach was initiated but aborted due to inability to puncture the radial artery were not included in the study. Enrolled patients were also excluded if the angiogram was performed solely via the femoral artery.
Groups:
- Terumo Control; Terumo Fast Release: A transparent unilateral compression device secured to the wrist via strap with velcro that was removed 1 hour after final deflation.
- Clo-Sur P.A.D.: A hydrophilic dressing with a high affinity for water and absorbs and controls body fluid that was removed on post-CATH day 1
Period: Overall Study
Arm/Group | Terumo Control | Terumo Fast Release | Clo-Sur P.A.D.
Started | 25 | 25 | 25
Completed | 15 | 20 | 18
Not Completed | 10 | 5 | 7

BASELINE CHARACTERISTICS:
Groups:
- Terumo Fast Release: A transparent unilateral compression device secured to the wrist via strap with velcro that was removed 15 minutes after final deflation.
- Total: Total of all reporting groups
Arm/Group | Terumo Control | Terumo Fast Release | Clo-Sur P.A.D. | Total
Number analyzed (Participants) | 25 | 25 | 25 | 75
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.4 (11.2) | 62.1 (8.3) | 64.1 (10.6) | 63.2 (10)
Age, Customized [Number; unit: participants]
  >=18 years | 25 | 25 | 25 | 75
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 3 | 11
  Male | 21 | 21 | 22 | 64
Region of Enrollment [Number; unit: participants]
  Canada | 25 | 25 | 25 | 75

OUTCOME MEASURES:

1. Primary Outcome: Bleeding Requiring Intervention After Initial Hemostasis Achieved
Description: Number of Participants with Bleeding Requiring Intervention after initial hemostasis achieved
Time Frame: Assessed after initial hemostasis achieved
Measure: Number; unit: participants
Arm/Group | Terumo Control | Terumo Fast Release | Clo-Sur P.A.D.
Number analyzed (Participants) | 25 | 25 | 25
participants | 2 | 6 | 3
Statistical Analysis 1: Comparison: Terumo Control vs Terumo Fast Release vs Clo-Sur P.A.D; Lancaster et. al. (2004) quoted the number 30 as a general sample size for a pilot study. Each arm of this study had 25 people (due to time constraints), giving a total of 75 people. The data were analyzed using t-tests for equality of means, a two-way analysis of variance (ANOVA), and chi-square. Significance was set at p < 0.05; Test type: Superiority or Other; p = 0.25, Chi-squared

2. Primary Outcome: Bleeding Requiring Intervention Post-CATH Day 1
Description: Number of Participants with Bleeding Requiring Intervention post-CATH Day 1
Time Frame: Assessed post-CATH Day 1
Population: Lancaster et. al. (2004) quoted the number 30 as a general sample size for a pilot study. Each arm of this study had 25 people (due to time constraints), giving a total of 75 people. The data were analyzed using t-tests for equality of means, a two-way analysis of variance (ANOVA), and chi-square. Significance was set at p < 0.05.
Measure: Number; unit: participants
Arm/Group | Terumo Control | Terumo Fast Release | Clo-Sur P.A.D.
Number analyzed (Participants) | 15 | 20 | 18
participants | 0 | 1 | 0
Statistical Analysis 1: Comparison: Terumo Control vs Terumo Fast Release vs Clo-Sur P.A.D; Test type: Superiority or Other; p = 0.47, Chi-squared

3. Secondary Outcome: Time to Discharge
Description: Time to discharge in minutes.
Time Frame: Assessed on day of angiogram.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Terumo Control | Terumo Fast Release | Clo-Sur P.A.D.
Number analyzed (Participants) | 25 | 25 | 25
minutes | 178.2 (50.4) | 134 (45.8) | 113.7 (48.0)
Statistical Analysis 1: Comparison: Terumo Control vs Terumo Fast Release; Test type: Superiority or Other; p = 0.002, ANOVA
Statistical Analysis 2: Comparison: Terumo Control vs Clo-Sur P.A.D; Test type: Superiority or Other; p < 0.001, ANOVA
Statistical Analysis 3: Comparison: Terumo Fast Release vs Clo-Sur P.A.D; Test type: Superiority or Other; p = 0.144, ANOVA

4. Secondary Outcome: Hematoma or Bruising at Discharge
Description: Number of Participants with hematoma or bruising at discharge
Time Frame: Assessed at discharge
Measure: Number; unit: participants
Arm/Group | Terumo Control | Terumo Fast Release | Clo-Sur P.A.D.
Number analyzed (Participants) | 25 | 25 | 25
participants | 1 | 2 | 0
Statistical Analysis 1: Comparison: Terumo Control vs Terumo Fast Release vs Clo-Sur P.A.D; Test type: Superiority or Other; p = 0.372, ANOVA

5. Secondary Outcome: Hematoma or Bruising Post-CATH Day 1
Description: Number of Participants with hematoma or bruising post-CATH Day 1
Time Frame: Assessed post-CATH day 1.
Measure: Number; unit: participants
Arm/Group | Terumo Control | Terumo Fast Release | Clo-Sur P.A.D.
Number analyzed (Participants) | 14 | 18 | 17
participants | 4 | 4 | 7
Statistical Analysis 1: Comparison: Terumo Control vs Terumo Fast Release vs Clo-Sur P.A.D; Test type: Superiority or Other; p = 0.468, Chi-squared

6. Secondary Outcome: Radial Artery Occlusion Post-CATH
Description: Number of Participants with Radial Artery Occlusion post-CATH
Time Frame: Assessed via plethysmography and palpation post-CATH
Measure: Number; unit: participants
Arm/Group | Terumo Control | Terumo Fast Release | Clo-Sur P.A.D.
Number analyzed (Participants) | 25 | 25 | 25
participants | 0 | 0 | 0

7. Secondary Outcome: Radial Artery Occlusion Post-CATH Day 1
Description: Number of Participants with Radial Artery Occlusion post-CATH Day 1
Time Frame: Assessed via plethysmography and palpation post-CATH day 1.
Measure: Number; unit: participants
Arm/Group | Terumo Control | Terumo Fast Release | Clo-Sur P.A.D.
Number analyzed (Participants) | 15 | 20 | 18
participants | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 2 days
Arm/Group | Terumo Control | Terumo Fast Release | Clo-Sur P.A.D.
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25 | 0/25

LIMITATIONS AND CAVEATS:
This was a pilot study. Not all extraneous variables were previously identified. The trial took place at a single-centre with a select number of cardiologists and nurses.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No